CLINICAL TRIAL: NCT06612307
Title: Sensitivity and Specificity of Leucocytes Subpopulation Versus Platelet Indices in Prediction of Clinical Outcome for Candidates With Sepsis. A Bi-centric Clinical Trial
Brief Title: Sensitivity and Specificity of Leucocytes Subpopulation Versus Platelet Indices in Prediction of Clinical Outcome for Candidates With Sepsis. A Bi-centric Observational Clinical Trial
Status: Not yet recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Ass professor anesthesia and pain, Minia University
Other Study IDs: Anet 19-2
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Leucocyte subpopulation and platelet indices analysis can predict clinical outcome

ELIGIBILITY:
Inclusion Criteria:

* Adult population of both sex, aged 20 or older admitted to the ICU with a diagnosis of sepsis were screened for inclusion within 48 h of presentation to the hospital. Sepsis was defined as per the Sepsis-3 definition, 6 ie, the presence of suspected or documented infection with organ dysfunction determined by an acute increase of sequential organ failure assessment (SOFA) score by 2 or more points

Exclusion Criteria:

* Patient refusal.
* History of surgery in the last 7 days from admission.
* Immunocompromised population ( post-transplantation, steroid use > 5 mg per day, malignancy, HIV, on chemotherapy).
* Population with history of thrombocytopenia ( ITP, aplastic anemia, drug induced)
* History of thrombocytosis ( idiopathic thrombocytosis, post-splenectomy)
* History of platelet transfusion one week before admission.
* Bone marrow transplanted population .
* Chronic liver and kidney disease.
* Von-Willebrand disease.
* Patients on antiplatelet therapy ( Aspirin, clopidogrel).
* Thrombocytopenic population ( ITP, TTP,HELLP) .
* Myelodysplastic or proliferative patients.
* Blood dyscarsiasis
* Obestetric parturients.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population admitted to the ICU with a diagnosis of sepsis were screened for inclusion within 48 h of presentation to the hospital. Sepsis was defined as per the Sepsis-3 definition, 6 ie, the presence of suspected or documented infection with organ dysfunction determined by an acute increase of sequential organ failure assessment (SOFA) score by 2 or more points
Sampling Method: Probability Sample
Enrollment: 161 (Estimated)
Dates: Start 2024-09-25 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of either leucocyte subpopulation, platelet indices with early clinical outcome | 1 week
  Post hoc analysis .... < 50 %= poor sensitivity..... > 50%= strong sensitivity
Specificity of either leucocyte subpopulation, platelet indices with early clinical outcome | 1 week
  Post hoc analysis .... < 50 %= poor sensitivity..... > 50%= strong sensitivity

SECONDARY OUTCOMES:
correlation between leucocytes at enrollment , 7 days with ICU mortality | 1 week
correlation between platelet indices at enrollment , 7 days with ICU mortality | one week
correlation between platelet indices at enrollment , 7 days with incidence of mechanical ventilation | 1 week
correlation between leucocytes at enrollment , 7 days with incidence of mechanical ventilation | 1week
correlation between leucocytes at enrollment , 7 days with incidence of acute kidney injury | 1 week
correlation between platelet indices at enrollment , 7 days with incidence of acute kidney injury | 1 week